CLINICAL TRIAL: NCT06695169
Title: Comprehensive Evaluation of the Integrated Smart Pump-EHR Technology in Eight Adult Acute and Intensive Care Units: A Mixed Method Study
Brief Title: Evaluation of the Integrated Smart Pump-EHR Technology in Eight Adult Acute and Intensive Care Units
Status: Recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY00000585
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Nurse's Role
Keywords: Integrated smart pumps; Integrated technology; Chart review

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nurses in ICU or Acute Care who administer medications using Smart infusion pumps: (A) Nurses from 8 acute and intensive care units (659 nurses total) will be invited to complete a survey about using the pumps.
  (B) Of these 659 nurses, 48 will join focus groups to share detailed thoughts on pump use.
  (C) Another 48 nurses will practice using the pumps in a simulation setting.
  The study will also review 200 patient records to check for any differences in documentation errors of IV medication volumes when using pump-EHR integration versus manually programming the pumps. Additionally, the study will analyze pump data from the last 6 months to see how often the technology is used and what types of alerts and programming errors occur. Furthermore, 20 healthcare team members will participate in interviews to understand the barriers and facilitators of technology use.

SUMMARY:
This study looks at the effects of using "smart pumps" that connect with the Electronic Health Record (EHR) in 8 adult ICU units.

We will interview nurses and healthcare team members to learn about any challenges with this technology.

All nurses in these units will be invited to complete a survey on how easy the technology is to use.

Some nurses will practice giving medications to "mannequins" in a simulation lab to see how they work with the pumps.

We will also look at existing data to find out how many nurses use the technology and what types of alerts or errors come up.

Finally, we will review patient charts to see if using the technology has increased or decreased errors in recording IV medication amounts.

DETAILED DESCRIPTION:
This mixed-methods design study focuses on understanding the complexity and consequences of implementing the integrated smart pumps-EHR technology in 8 adult acute and intensive care units (ICUs) using a comprehensive evaluation approach. The evaluation will include (1) analyzing use manifestations in terms of nurse adoption, alarms, alerts, and error messages associated with technology use, (2) examining the usability of the integrated technology, and (3) identifying influential factors that facilitate or hinder technology adoption.

ELIGIBILITY:
Inclusion Criteria:

* Research Aims 1 (adoption rate) and 2 (frequency and types of alerts and programming error ). We will include all IV medications and fluids delivered via smart infusion pumps within the past 6 months. We anticipate the dataset to include more than 180,000 of medications and fluid administration events.
* Research Aim 3 (documentation errors ). We will select 200 IV medications that were administered with solutions using chart audit. To be included, the selected IV medications should be diluted with at least 100 ml solution. The choice of the 100 ml cutoff point was based on it being the minimum volume for the majority of IV medication administrations.
* Research Aims 4, 5, 6, and 7 (usability of the technology, nurse perception, predictors of nurse perception, nurse experience with technology). Eligibility criteria will be confined to registered nurses with at least an associate degree in nursing.
* Research Aim 8 (multidisciplinary team experience with technology). The inclusion criteria for the group of multidisciplinary representatives encompass participation in pump implementation and pumps-related quality improvement initiatives.

Exclusion Criteria:

* Research Aims 1 and 2. Bolus medications will be excluded due to the distinct workflow associated with their administration.
* Research Aim 3. Medications with solution volumes lower than 100 ml will be excluded.
* Research Aims 4, 5, 6, and 7. Licensed vocational nurses (LVN) and licensed practical nurses (LPN) will be excluded due to their non-involvement in IV medication administration. Additionally, and for Research Aim # 7, the group of 48 nurses who will engage in the usability testing will not be part of the focus group interviews to ensure a broader participation among nurses.
* Research Aim 8: Stakeholders from the different hospital's departments and councils (e.g., nursing, biomedical engineering, pharmacy, risk and management, technology committees, etc.) who were not part of the implementation process of infusion pumps in 2018 and 2020 or are not involved in continuous quality initiatives related to infusion pump adoption and quality measures tracking will be excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nurses who use integrated smart pump technology to administer IV drugs and fluids will take part in interviews, simulations, and surveys.
  Additionally, a sample of multidisciplinary team members involved in the implementation of smart pumps in 2018, the integration of smart pumps with the electronic health record in 2020, or past/current pump-related quality improvement initiatives will participate in interviews.
Sampling Method: Non-Probability Sample
Enrollment: 659 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Pump adoption rate | 6 months
  Data from the pumps over the past 6 months will be reviewed and analyzed to understand how often nurses use the integrated pump-EHR (or electronic health record) technology versus manually programming the pumps when administering medications. Z-test will be used to test the difference in percentage in adoption rate.
Alerts messages | 6 months
  Data from the pumps over the past 6 months will be reviewed to examine the difference in frequency of alert messages (including programming error messages) generated when manually programming the pump versus using the pump-EHR integrated technology. Data will be analyzed using chi-square.
Errors in documenting the volume of IV medications | 4 months
  200 patient charts will be reviewed to compare documentation errors in IV medication volumes when using pump-EHR integration versus manual pump programming.

SECONDARY OUTCOMES:
Usability of the Pumps | 9 months
  During observations of 48 nurses' interactions with the pumps in a simulated environment, we will identify the navigation paths nurses follow to program the pumps (through recording of nurse-pump navigation), examine usability errors (through recording of nurse-pump navigation), record the time taken by nurses to navigate the pumps to administer IV medications (through recording of nurse-pump navigation), assess perceived workload during pump navigation (using a survey), and assess nurse experience and perceived challenges during task completion (using the debriefing session).
Nurse perception of the usability of the integrated smart pump technology | 6 months
  We will send a survey to all nurses who work in the 8 acute and intensive care units to understand their perceptions about the technology. Descriptive statistics will be used to analyze the results.
Factors that facilitate or hinder technology adoption | 11 months
  We will use semi-structured interviews to explore bedside nurses' experiences with the integrated smart pump-EHR technology, including any challenges they face.
  Additionally, we will interview a multidisciplinary healthcare team to understand the organizational and contextual factors that help or hinder the adoption of this technology.
  All interviews will be transcribed by professionals from Rev, a transcription vendor. Data will be entered into nVivo software. The 4-stage content analysis methodology by Bengtsson (2016) will be used to categorize narrative data into themes.

CONTACTS AND LOCATIONS:
Overall Officials: Azizeh Sowan, PhD, RN, MSN, MSDA, MBA, FAAN, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University Health, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
The specific individual participant data (IPD) that will be shared will be limited to quantitative data. These will include the de-identified responses to the survey, the log data retrieved from smart pumps, and the de-identified results of the chart audit.
Time Frame: The IPD will be available starting 6 months after the publication of the study results. The data will remain available for a period of 5 years from the end date of data collection.
Access Criteria: The de-identified IPD will be made available to researchers upon reasonable request for purposes of secondary analysis or meta-analysis only. Access will be granted to qualified researchers affiliated with academic, non-profit, or government institutions who provide a detailed research proposal outlining their objectives and methods.
  Researchers will need to sign a data use agreement that outlines the terms of access, including proper data handling, acknowledgment of the original study, and compliance with ethical standards. The data will be shared electronically via a secure data-sharing platform, and access will be time-limited based on the approved use.
  For the URL below, No dedicated webpage is available at this time. For more information about the IPD sharing plan, interested researchers may contact [Azizeh Sowan, Sowan@uthscsa.edu and Ana Vera, ana.vera@uhtx.com]